CLINICAL TRIAL: NCT06238271
Title: Evaluation of the Long-term Efficacy and Safety of Monofocal Plate Haptic Intraocular Lens to be Implanted Into the Eye in Patients Undergoing Cataract Surgery
Brief Title: Evaluation of the Long-term Efficacy and Safety of Monofocal Plate Haptic Intraocular Lens
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuzuncu Yil University (Other)
Collaborators: VSY Biotechnology (Unknown)
Responsible Party: Principal Investigator, Erbil Seven, MD, Associate Professor, Yuzuncu Yil University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 02
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Lens Implantation, Intraocular; Cataract
Keywords: Cataract; Intraocular lens implantation; Phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- UDM 611 (Experimental): Acriva BB UDM 611 intraocular lens will be implanted into the capsular bag in patients who undergo cataract extraction with phacoemulsification.
  Interventions: Device: Acriva BB UDM 611

INTERVENTIONS:
Device: Acriva BB UDM 611 — Acriva BB UDM 611 intraocular lens will be implanted into the capsular bag in patients who undergo cataract extraction with phacoemulsification.

SUMMARY:
Our study aims to determine the efficacy and safety of the monofocal plate haptic intraocular lens to be implanted in patients planning for cataract surgery and to determine the complications that may develop due to the lens.

DETAILED DESCRIPTION:
This study was planned to be performed on 300 eyes with surgical indication due to cataracts in Van Yüzüncü Yıl University Faculty of Medicine Ophthalmology Outpatient Clinic. Uncorrected and best-corrected visual acuity, subjective refraction, slit-light biomicroscopy, optical biometry, anterior segment optical coherence tomography, intraocular pressure, endothelial cell count in the pre-and postoperative (1st, 3rd, and 12th months) controls of the patients. Fundus examination will be performed, and postoperative complications and accompanying ocular pathologies will be recorded. Data before and after surgery effectiveness will be evaluated. Reliability will be interpreted by considering postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient informed of the consequences and constraints of the protocol and who has given his/her written informed consent;
* Patients of any gender
* Assured follow-up examinations
* Biometry measurement preferably compatible with the Lenstar evaluation;
* IOL implanted into the capsular bag with IOL model Acriva BB UDM 611 (UVE material) in one or both eyes

Exclusion Criteria:

* BCVA not available preoperatively or better than 0.3 logMAR pre-op
* Patients unable to meet the limitations of the protocol or likely to non-cooperation during the trial
* Patients with peroperative complications (Such as capsulorhexis problems that affect centralization, failure of the IOL implanting into the bag, posterior capsular rupture, iris damage, vitreous loss, IOL damage, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 12 to 18 months after surgery
  Monocular best corrected distance visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yil University, Van, Turkey (Türkiye)